CLINICAL TRIAL: NCT01301391
Title: Phase II Study Of Oral PHA-848125AC In Patients With Malignant Thymoma Previously Treated With Multiple Lines Of Chemotherapy
Brief Title: Study Of Oral PHA-848125AC In Patients With Malignant Thymoma Previously Treated With Multiple Lines Of Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For the last patient still on treated nominal therapeutic use of the Milciclib was approved at INT Milano.
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDKO-125a-007
Record Dates: First submitted 2011-02-15; First posted 2011-02-23 (Estimated); Results first posted 2018-10-04 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Malignant Thymoma
Keywords: B3 and C malignant thymoma
MeSH Terms: conditions — Thymoma | interventions — N,1,4,4-tetramethyl-8-((4-(4-methylpiperazin-1-yl)phenyl)amino)-4,5-dihydro-1H-pyrazolo(4,3-h)quinazoline-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milciclib (Experimental): Milciclib Maleate capsules
  Interventions: Drug: Milciclib Maleate

INTERVENTIONS:
Drug: Milciclib Maleate — 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Number of cycles: until disease progression or unacceptable toxicity.
  Other Names: PHA-848125AC

SUMMARY:
The intent of the study is to assess the antitumor activity of PHA-848125AC in patients with recurrent or metastatic, unresectable malignant thymoma previously treated with multiple lines of chemotherapy.

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, phase II clinical trial design with an early stopping rules. PHA-848125AC will be administered to patients with recurrent metastatic unresectable B3 thymoma or thymic carcinoma who have received more than one line of prior systemic therapy for advanced / metastatic disease. The intent of the study is to assess the antitumor activity of PHA-848125AC and ultimately to improve the outcome of the patients. The primary end point for this study is a progression free survival rate of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated IRB/Approved Informed Consent
* Histologically or cytologically proven diagnosis of unresectable B3 thymoma or thymic carcinoma recurrent or progressing after more than one prior systemic therapy for advanced / metastatic disease
* Presence of measurable disease
* Age >=18 years old
* ECOG performance status 0-1
* Negative pregnancy test (if female in reproductive years)
* Use of effective contraceptive methods if men and women of child producing potential
* Adequate liver function Total Serum Bilirubin <=1.5 x upper limit of normal (ULN) Transaminases (AST/ALT) <=2.5ULN (if liver metastases are present, then <=5ULN is allowed) ALP <=2.5ULN (if liver and/or bone metastases are present, then <=5ULN is allowed)
* Adequate renal function Serum Creatinine <=ULN or Creatinine Clearance calculated by Cockcroft and Gault's formula > 60 mL/min
* Adequate hematologic status ANC >=1,500cells/mm3 Platelet Count >= 100,000cells/mm3 Hemoglobin >=9.0g/dL
* Two weeks must have elapsed since completion of prior chemotherapy, minor surgery, radiotherapy (provided that no more than 25% of bone marrow reserve has been irradiated)
* Resolution of all acute toxic effects of any prior treatments to NCI CTC (Version 3.0) grade <=1

Exclusion Criteria:

* Any of the following in the past 6 months: myocardial infarction, uncontrolled cardiac arrhythmia, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis
* Grade >1 retinopathy
* Known brain metastases
* Known active infections
* Pregnant or breast feeding women
* Diabetes mellitus uncontrolled
* Gastrointestinal disease that would impact on drug absorption
* Patients under treatment with anticoagulants or with coagulation disorders or with signs of hemorrhage at baseline
* Patients with previous history or current presence of neurological disorders (with the exception of myasthenia gravis), including epilepsy (although controlled by anticonvulsant therapy), Parkinson's disease and extra-pyramidal syndromes.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, MD., Principal Investigator — National Cancer Institute (NCI); Marina C. Garassino, MD., Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano; Giuseppe Giaccone, MD, Principal Investigator — MedStar Gergetown University Hospital
Locations (3):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - NIH, Center for Cancer Research, Medical Oncology, Bethesda, Maryland
- Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, (mi), Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 02 Feb 2011 to 28 Jan 2016 by 2 centers in US and one in Italy.
Pre-assignment Details: Four patients were screening failure.
Groups:
- Milciclib: Milciclib Maleate capsules
  Milciclib Maleate: 150 mg/day once daily, for 7 consecutive days (days 1 to 7) followed by 7 days of rest (days 8 to 14) in a 2-week cycle.
  Number of cycles: until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Milciclib
Started | 30 (On treatment until disease progression, patient withdrawal of consent, or unacceptable toxicity.)
Completed (Follow up for survival: up to the end of study or for no more than 2 years from end of treatment.) | 4
Not Completed | 26
Not completed — Death | 13
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2
Not completed — Sponsor's decision | 8

BASELINE CHARACTERISTICS:
Arm/Group | Milciclib
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  Black | 2
  Asian | 3
  Not Listed | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
  Italy | 15
World Health Organization classification (International Classification of Diseases) [Count of Participants; unit: Participants]
  B3 - Well Differentiated Thymic Carcinoma | 17
  C - Thymic Carcinoma | 13
Tumor extent at study entry [Count of Participants; unit: Participants]
  Metastatic | 30
  In situ | 0
Masaoka clinical staging at study entry [Count of Participants; unit: Participants] — Staging used to evaluate invasiveness of the tumor.
  Participants
    Stage I: Grossly and microscopically encapsulate | 0
    Stage II: Thymoma invades beyond the capsule | 0
    Stage III: Macroscopic invasion neighboring organs | 0
    Stage IVA: Pleural or pericardial dissemination | 7
    Stage IVB: Hematogenous or lymphatic dissemination | 10
    Not assessed | 6
    Not available | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 3 Months
Description: The proportion of successes (i.e. patients alive and progression-free at 3 months since treatment start) out of the total number of evaluable patients.
Time Frame: 3 months since treatment start
Population: Evaluable patients, i.e., consists of all eligible and treated patients who fulfill the following additional conditions: 1) they receive at least 80% of drug in the first two cycles overall; 2) they have baseline and > or = 1 on-treatment tumor/oncologic assessment(s) or die before tumor re-assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Milciclib
Number analyzed (Participants) | 24
Participants
  Success | 13
  Failure | 11
Statistical Analysis 1: Comparison: Milciclib; H0:p≤ 25% vs H1:p> 25% with an interesting PFS-3 rate of 50% (median PFS of 3 months), alpha=0.05 and beta=0.10, 30 evaluable patients are required for a single stage trial. If at the end of the trial 12 or more out of 30 evaluable patients are alive and progression-free at 3 months since the treatment start date, the null hypothesis are rejected. A Fleming multiple-testing procedure is applied. If >=4 successes out of the first 15 patients are observed, accrual will continue up to 30; Test type: Superiority; p < 0.001, Fisher Exact — A priori threshold for statistical significance = 0.05; Single proportion = 0.54, 95% CI 2-sided [0.33 to 0.74]

2. Secondary Outcome: Adverse Events (NCI CTCAE) and Hematological and Blood Chemistry Parameters
Description: The adverse events (AEs) were coded with the Medical Dictionary for Regulatory Activities (MedDRA) and their severity graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The following subsets of AEs were considered: serious AEs, AEs with CTCAE grade 3-5, AEs with a relationship to study treatment classified by the Investigator as possible or probable or definite and AEs reported as leading to discontinuation from treatment.
  Laboratory test values were graded according to the NCI CTCAE scale, v3.0, whenever possible. For each laboratory test included in the NCI CTCAE system, the incidence of abnormalities were evaluated by considering the worst occurrence for each patient throughout the whole treatment period.
Time Frame: Adverse events: from date treatment consent signed to 28 days after last treatment; hematology/blood chemistry tests: at baseline and between Day 11-14 of each cycle of a maximum total of 48 two-week cycles.
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Milciclib
Number analyzed (Participants) | 30
Participants
  N° patients with Adverse Events | 30
  N° patients with abnormal Hematology test | 28
  N° patients with abnormal Blood chemistry test | 27

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Point and 95% confidence interval estimates was calculated for the objective tumor response rate (confirmed CRs or PRs). The determination of antitumor efficacy was based on objective tumor assessments made according to the RECIST guideline (version 1.1). The analysis was performed in the evaluable population.
Time Frame: Assessments were made every 6 weeks from start date until PD or up to a maximum duration of 134 weeks.
Population: Evaluable population: the patient population consists of all eligible and treated patients who fulfill the following additional conditions: 1) they receive at least 80% of drug in the first two cycles overall; 2) they have baseline and > or = 1 on-treatment tumor/oncologic assessment(s) or die before tumor re-assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Milciclib
Number analyzed (Participants) | 24
Percentage of patients | 4.2 [0.11 to 21.12]

4. Secondary Outcome: Disease Control Rate (ORR+SD Rate)
Description: Point and 95% confidence interval estimates was calculated for the disease control rate (confirmed CRs / PRs and SD > or = 6 weeks). The analysis was performed in the evaluable patient populations.
Time Frame: Assessments were made every 6 weeks from start date until PD or up to a maximum duration of 134 weeks.
Population: Evaluable patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Milciclib
Number analyzed (Participants) | 24
Percentage of patients | 83.3 [62.62 to 95.26]

5. Secondary Outcome: Duration of Response
Description: Calculated in patients achieving a confirmed objective tumor response by RECIST version 1.1 criteria.
Time Frame: Assessments were made every 6 weeks from start date until PD or up to a maximum duration of 134 weeks.
Population: Patients achieving a confirmed objective tumor response by RECIST version 1.1 criteria.
Measure: Number; unit: Months
Arm/Group | Milciclib
Number analyzed (Participants) | 1
Months | 2.76

6. Secondary Outcome: Overall Survival
Description: The length of time from either the date of diagnosis or the start of treatment for a disease, such as cancer, and to the date in which the patients diagnosed with the disease are still alive. Kaplan-Meier estimates as percentage of patients alive.
Time Frame: Every 6 weeks during Follow-Up until PD or new therapy start; every 6 months thereafter, up to 2 years from the last dose of study drug.
Population: Evaluable patients
Measure: Number; unit: percentage of patients dead at 21 months
Arm/Group | Milciclib
Number analyzed (Participants) | 24
percentage of patients dead at 21 months | 41.666

7. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse. In a clinical trial, measuring the progression-free survival is one way to see how well a new treatment works.
Time Frame: Assessments were made every 6 weeks from start date until PD or up to a maximum duration of 134 weeks.
Population: Evaluable patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Milciclib
Number analyzed (Participants) | 24
Months | 9.76 [4.11 to 17.45]

ADVERSE EVENTS:
Time Frame: Adverse events were reported for patients from consent signed to 28 days after last dose of study drug. Individual patient adverse event reporting ranged from 5.1 weeks to 141.3 weeks with a median of 19.28 weeks.
Arm/Group | Milciclib
All-Cause Mortality (participants affected / at risk) | 13/30
Serious Adverse Events (participants affected / at risk) | 14/30
Other Adverse Events (participants affected / at risk) | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milciclib (N=30)
Haemoptisys (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain NOS (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction NOS (Gastrointestinal disorders) | 1 (1)
Pneumonia NOS (Infections and infestations) | 2 (2)
Sepsis NOS (Infections and infestations) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating increased (Skin and subcutaneous tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase NOS increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Epididymitis NOS (Reproductive system and breast disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milciclib (N=30)
Nausea (Gastrointestinal disorders) | 25 (92)
Diarrhoea NOS (Gastrointestinal disorders) | 18 (70)
Vomiting NOS (Gastrointestinal disorders) | 17 (66)
Constipation (Gastrointestinal disorders) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Abdominal pain NOS (Gastrointestinal disorders) | 2 (4)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder NOS (Gastrointestinal disorders) | 2 (4)
Asthenia (General disorders) | 11 (22)
Fatigue (General disorders) | 11 (17)
Pyrexia (General disorders) | 7 (9)
Oedema peripheral (General disorders) | 5 (5)
Chest pain (General disorders) | 3 (3)
Pain NOS (General disorders) | 2 (4)
Pain exacerbated (General disorders) | 2 (2)
Tremor (Nervous system disorders) | 11 (30)
Dizziness (Nervous system disorders) | 7 (12)
Paraesthesia (Nervous system disorders) | 4 (5)
Dysgeusia (Nervous system disorders) | 3 (3)
Haedache (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 8 (8)
Appetite decreased NOS (Metabolism and nutrition disorders) | 2 (3)
Dehydratation (Metabolism and nutrition disorders) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (4)
Lipase increased (Investigations) | 4 (11)
Alanine aminotransferase increased (Investigations) | 3 (5)
Blood amylase increased (Investigations) | 3 (6)
Weight decreased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (7)
Conjunctivitis (Eye disorders) | 2 (3)
Ocular discomfort (Eye disorders) | 2 (2)
Photopsia (Eye disorders) | 2 (3)
Influenza (Infections and infestations) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (3)
Azotaemia (Renal and urinary disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT01301391/Prot_000.pdf
  • Statistical Analysis Plan: CDKO-125a-007_ALG_V1 (2013-04-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT01301391/SAP_001.pdf
  • Statistical Analysis Plan: CDKO-125a-007_TLG_V1 (2013-04-22): https://cdn.clinicaltrials.gov/large-docs/91/NCT01301391/SAP_002.pdf